CLINICAL TRIAL: NCT06851390
Title: Inflammation and Cerebral Oxygenation in Preterm Newborns Following Fetal Red Blood Cell Transfusion Compared to Adult Red Blood Cell Transfusion
Acronym: INCONTRA
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Stefano Ghirardello, MD, Chief of Neonatal Unit and Neonatal Intensive care Unit, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: INCONTRA
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Preterm Newborns
Keywords: preterm newborn; packed RBC; inflammation markers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preterm newborns undergoing cord/placental RBC transfusion
- preterm newborns undergoing adult RBC transfusion

SUMMARY:
Among diseases associated with premature birth, retinopathy of prematurity (ROP) is one of the most important causes of childhood blindness. ROP develops in the immature retina as a consequence of prolonged exposure to hyperoxia. A body of evidence suggests a connection between ROP and the number of red blood cell (RBC) transfusions. Moreover, in newborns receiving repeated transfusions, fetal hemoglobin (HbF) progressively declines. Our NICU participate to the BORN (umBilical blOod to tRansfuse preterm Neonates) trial, a double-blind, multi-center, randomized controlled trial with the aim of evaluating if preterm newborns randomized to receive cord blood (CB)-transfusions have a lower incidence of ROP, compared to newborns transfused with adult RBC cells. In the context of BORN trial, with this ancillary INCONTRA study, the investigators aim to explore the inflammatory burden, potentially impacting on development of the preterm newborn comorbidities, following CB-RBC transfusions, compared to adult RBC transfusions. to estimate the change in pro-inflammatory cytokine (IL-1β, IL-8, TNF-α) and MCP-1, MIF, s-ICAM levels levels circulating in preterm newborns before and after transfusion, Moreover, we want to monitor cerebral oxygenation and oxygenation delivery to the brain during and after the transfusion of the two different RBC products. Moreover, the investigators aim to monitor cerebral oxygenation and oxygenation delivery to the brain during and after the transfusion of the two different RBC products.

ELIGIBILITY:
Inclusion criteria:

* gestational age (GA) at birth < 28 weeks
* signed informed consent of parents.

Exclusion criteria:

* maternal-fetal immunization, hydrops fetalis
* major congenital malformations associated or not with genetic syndromes
* previous transfusions
* hemorrhage at birth requiring transfusion (within 12 hours from birth)
* congenital viral infections
* outborn infants who received RBC transfusions before admission to the Neonatal Intensive Care Units participating to the study
* health care team deeming it inappropriate to approach the infant's family for informed consent
* Severe IgA deficiency
* Any life-threatening comorbidity or any other medical condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion.

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Our NICU participate to the multicenter trial, BORN (umBilical blOod to tRansfuse preterm Neonates) enrolling newborns randomized to receive cord blood or adult transfusions. They were also evaluated in the present monocentric ancillary study (INCONTRA) to measure newborn's plasma concentration of inflammation markers
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
measure of pro-inflammatory cytokine levels (IL-1β, IL-8, TNF-α) andMCP-1, MIF, s-ICAM levelscirculating in preterm newborns before transfusion and two hours after transfusion | During the first 4 months of life.

SECONDARY OUTCOMES:
trend of cerebral rStO2, measured by near infrared spectroscopy (NIRS) | In the time of time of transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
A decision has not been made yet